CLINICAL TRIAL: NCT04603534
Title: Empathy and Attitude Upon An Aged Body: Aged Simulation Suit Among Undergraduate Physiotherapy Students
Brief Title: Aged Simulation Suit Among Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Head of Geriatric Rehabilitation Department, Izmir Bakircay University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/14
Record Dates: First submitted 2020-10-15; First posted 2020-10-27 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Empathy; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Other: Aged Simulation Suit

INTERVENTIONS:
Other: Aged Simulation Suit — The aged simulation suit (Sakamoto Model M716, Tokyo, Japan) will be worn by students. The simulation suit consist of a several items such as loads, a soft material band with Velcro, glasses, ear plugs, gloves, belts and a cane. All the items are need to simulate one's posture just like in elderly person. Small, medium and large sizes of suits are provided by the company thereby each suit is suitable for each student related to their wearing size. Prior to this study, a total of three sets of suits will be gathered. Then, each student will perform each pre-defined scenarios step by step after the suit is worn. During the activities no help or leading will be given to the students. However, one of the researchers will supervise the students during the activities so that to integrate a safe platform. In addition, each student will be informed that if he/she can terminate the activity whenever it is required.

SUMMARY:
Turkey is the second fastest aging country in the world. According to the Turkey Statistical Institute's data, the distribution of the population aged 65 and over is expected to be 25.6% in 2080. Today, studies have been started to determine the empathy and attitudes of the young generation, especially the younger generation, towards older individuals and to develop them. In this context, it is thought that the simulation designed to simulate the aging process of human beings may have a positive effect on students' understanding of aging and perception of aging. In this study, the effect of aged simulation suit on empathy and attitudes towards elderly people will be determined in Physiotherapy and Rehabilitation undergraduate students.

DETAILED DESCRIPTION:
Attitude is defined as a positive or negative assessment of people, objects or events that reflect one's knowledge, emotions, and behavior towards people, objects or events. Physical degeneration in the elderly can easily lead to prejudice or discrimination against older adults, especially in the younger generation. The younger generation sees older adults as a different group and labels them with negative traits. However, education has an important role in changing attitudes towards older people and developing professional cultures. In this context, the positive attitudes and behaviors of healthcare professionals (doctors, nurses, physiotherapists, etc.) starting from the pre-graduation period are of great importance for quality health services.

Empathy, which consists of emotional, cognitive, operational, and physiological behavior and reaction compounds, was mostly evaluated as a process of relationships and attitudes. Healthcare providers should be able to grasp patients' perspectives (cognitive empathy) and relate to their emotions and experiences (emotional empathy). It can be difficult to understand other people's perspectives, especially if they have not experienced disability due to aging or disease. It has been reported in the literature that health professionals lack empathy and understanding towards older individuals. It has been suggested that empathy in patient care can be developed at a basic level and through vocational education. Defining the attitudes of healthcare professionals and students and implementing new educational strategies that encourage positive attitudes towards the elderly while they are still students are important for increasing the quality of healthcare offered to the elderly and developing a positive attitude.

In medical and health sciences undergraduate education, there has been a lack of specific lessons on which directly focuses empathy, yet simulation-based modalities have been shown to be impacted on students' perceptions regarding attitude and empathy.

Thus, this study aims to assess the attitude and empathy level toward on elderly people among health sciences undergraduate students. The intervention which is mainly based upon wearing an aged simulation suit through some activities related to independent living and mobility has been planned to performed.

ELIGIBILITY:
Inclusion Criteria:

* Being volunteer to participate

Exclusion Criteria:

* Having an advanced visual and balance problems especially associated with inner ear

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-03-15 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline The Jefferson Scale of Empathy Health Professions Students immediately after the intervention | At baseline and immediately after the intervention
  The Jefferson Scale of Empathy Health Professions Students (JSE-HPS) was originally developed by Jefferson University intended to measure empathy levels for health professionals. The JSE-HPS consists of a total 20-items each scored by seven point Likert Scale as 1: "Strongly disagree" through 7: "Strongly agree". 10 out of 20 items are scored directly according to the Likert weights while the other half are reversely scored. The minimum and maximum scores for JSE-HPS can be reached to 20 and 140, respectively. The more the higher scores indicate more empathic aspect or vice versa.
Change from Baseline Kogan's Attitude towards Old People scale immediately after the intervention | At baseline and immediately after the intervention
  The scale consists a total of 34 items which was originally developed by Kogan et al. The same as in JSE-HPS, seventeen items which are directly scored as Likert weights according to the 6 point Likert scale in which 1: "Strongly Disagree" through 6: "Strongly agree" while the rest of seventeen items are scored reversely. The minimum and maximum points of Kogan's Attitude towards Old People (KAOP) scale can be 34 and 238. The interpretation of score of KAOP scale is linear in which higher scores indicate a more positive attitude while lower scores indicate the worse. Reliability of the total KAOP scale were found in different studies as 0.87 and 0.89.

SECONDARY OUTCOMES:
Semi-structure Interview | Immediately after the intervention
  Experiences and emotions regarding the aged simulation suit will be collected from the students by asking reflective questions for each student one by one. Qualitative discussion will be made by taking experiences and perceptions of students upon the aged simulation suit.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided